CLINICAL TRIAL: NCT01163188
Title: Social Adjustment and Quality of Life After Very Preterm Birth: Risk and Resiliency From Infancy to Adulthood
Brief Title: Social Adjustment and Quality of Life After Very Preterm Birth
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Warwick (Other); Ludwig-Maximilians - University of Munich (Other); Bundesverband Bunter Kreis e.V. (Industry); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Peter Bartmann, Prof. Dr. Dr., University Hospital, Bonn
Other Study IDs: 01ER0801
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Low Birth Weight; Premature Birth
Keywords: very low birthweight/ very preterm children; Bavarian Longitudinal Study (BLS); Quality of life and social adjustment in adulthood
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — hair
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Proband: Very low birth weight children (< 32 weeks of gestation) and/ or Very preterm children (< 1500 g birthweight) of the Bavarian Longitudinal Study
- Controls: Term born children of the Bavarian Longitudinal Study

SUMMARY:
The major aim is the follow-up of the highest risk group (< 32 weeks gestation/ < 1500 birthweight) and their controls of the Bavarian Longitudinal Study (BLS) at the age of 24-27 years. The focus will be the identification of risk, protective and resiliency factors for cognitive and behavioural development and quality of life.

MRIs of the central nervous system will be conducted to examine aberrant activation patterns during the "attention network task" in stratified subgroups. Data driven MRI methods will be evaluated in relation to clinical, behavioural and developmental parameters.

DETAILED DESCRIPTION:
The major aim is the follow-up of the highest risk group (< 32 weeks gestation/ < 1500 birthweight) and their controls of the Bavarian Longitudinal Study (BLS) at the age of 24-27 years. All probands have been assessed previously, neonatally and at additional six time points, the last time at the age of 12-13 years. The focus will be the identification of risk, protective and resiliency factors for cognitive and behavioural development and quality of life. On the basis of previously assessed data statistical modelling of child development until age 8.5 years will be conducted across the total range of gestation from 26-42 weeks to identify social factors amenable to intervention which could be associated with a positive development especially in moderate prematurity. In addition, cross-validation of the findings is planned by means of comparisons with three international studies (Millenium Cohort, GB; POPS, NL; EPICure, GB). MRIs of the central nervous system will be conducted to examine aberrant activation patterns during the "attention network task" in stratified subgroups. Data driven MRI methods will be evaluated in relation to clinical, behavioural and developmental parameters. In line with the objectives of funding there will be a further follow-up of the BLS to answer important questions regarding health and development of very small preterms.

ELIGIBILITY:
Inclusion Criteria:

* very low birth weight VLBW (< 1500g birthweight)and/ or
* very preterm birth VPT (< 32 weeks of gestation)
* Members of the Bavarian Longitudinal Study

Exclusion Criteria:

* missing compliance

Ages: 24 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Very low birthweight (< 1500g birthweight) and/ or very preterm children (< 32 weeks of gestation) and a control group of term born children from the Bavarian Longitudinal Study
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 years
  Psychologic Interview, face-to-face in Adulthood on one day:
  Life Course Interview Wechsler Adult Intelligence Scale Diagnostic Expertsystem Interview for psychotic Symptoms Broad Autism Phenotype Questionaire DANVA Questionaire for ADHD Symptoms TRCB Health Utility Index London Handicap Scale WHO-Quality of Life Satisfaction with Life Scale ANT-I Task Additional Lenght, Weight, Head-, Waist-, Hipfcircumferende were measured. These examinations will be matched with these of previous examinations.
  At the second examinationday the selected probands who are physically and mentally able to undergo a functional MRI, will be examined with:
  structure-examination DTI Resting Brain ANT N-back These examination will be compared with literature data.

SECONDARY OUTCOMES:
Quality of life | 3 years
  At the psychological interview the testinstrumentes can be enlarged if possible:
  Rapid Automatized Naming Test Color -Word Interferencetest Regensburger verbal fluency test Visual Search and Attention Test Smily task Beck Depression Inventar Achenbach Young Adult Self Report Pittsburgh Sleep Quality index Warwick Edinburgh Mental Wellbeing Scale questionaire for generally health Rosenberg Skala self-esteem mass Arnett Inventory of Sensation Seeking Big Five Inventory-10

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bartmann, Prof., Principal Investigator — University of Bonn, Zentrum für Kinderheilkunde, Abt. Neonatologie; Dieter Wolke, Prof., Study Director — University of Warwick
Locations (1):
- Institut für Sozialmedizin in der Pädiatrie Augsburg, Augsburg, Bavaria, Germany

REFERENCES:
- [Background] Wolke D, Schmid G, Schreier A, Meyer R. Crying and feeding problems in infancy and cognitive outcome in preschool children born at risk: a prospective population study. J Dev Behav Pediatr. 2009 Jun;30(3):226-38. doi: 10.1097/DBP.0b013e3181a85973. PMID 19433987
- [Background] Schmid G, Schreier A, Meyer R, Wolke D. A prospective study on the persistence of infant crying, sleeping and feeding problems and preschool behaviour. Acta Paediatr. 2010 Feb;99(2):286-90. doi: 10.1111/j.1651-2227.2009.01572.x. Epub 2009 Nov 2. PMID 19886897
- [Background] Verrips E, Vogels T, Saigal S, Wolke D, Meyer R, Hoult L, Verloove-Vanhorick SP. Health-related quality of life for extremely low birth weight adolescents in Canada, Germany, and the Netherlands. Pediatrics. 2008 Sep;122(3):556-61. doi: 10.1542/peds.2007-1043. PMID 18762526
- [Result] Jaekel J, Baumann N, Wolke D. Effects of gestational age at birth on cognitive performance: a function of cognitive workload demands. PLoS One. 2013 May 24;8(5):e65219. doi: 10.1371/journal.pone.0065219. Print 2013. PMID 23717694
- [Result] Wolke D, Chernova J, Eryigit-Madzwamuse S, Samara M, Zwierzynska K, Petrou S. Self and parent perspectives on health-related quality of life of adolescents born very preterm. J Pediatr. 2013 Oct;163(4):1020-6.e2. doi: 10.1016/j.jpeds.2013.04.030. Epub 2013 May 30. PMID 23726545
- [Result] Johnson S, Wolke D. Behavioural outcomes and psychopathology during adolescence. Early Hum Dev. 2013 Apr;89(4):199-207. doi: 10.1016/j.earlhumdev.2013.01.014. Epub 2013 Feb 27. PMID 23455605
- [Result] Jaekel J, Wolke D, Bartmann P. Poor attention rather than hyperactivity/impulsivity predicts academic achievement in very preterm and full-term adolescents. Psychol Med. 2013 Jan;43(1):183-96. doi: 10.1017/S0033291712001031. Epub 2012 May 21. PMID 22608065
- [Result] Hall J, Wolke D. A comparison of prematurity and small for gestational age as risk factors for age 6-13 year emotional problems. Early Hum Dev. 2012 Oct;88(10):797-804. doi: 10.1016/j.earlhumdev.2012.05.005. Epub 2012 Jun 12. PMID 22698435
- [Result] Jaekel J, Wolke D, Chernova J. Mother and child behaviour in very preterm and term dyads at 6 and 8 years. Dev Med Child Neurol. 2012 Aug;54(8):716-23. doi: 10.1111/j.1469-8749.2012.04323.x. Epub 2012 May 24. PMID 22624879
- [Result] Heinonen K, Raikkonen K, Pesonen AK, Andersson S, Kajantie E, Eriksson JG, Wolke D, Lano A. Longitudinal study of smoking cessation before pregnancy and children's cognitive abilities at 56 months of age. Early Hum Dev. 2011 May;87(5):353-9. doi: 10.1016/j.earlhumdev.2011.02.002. Epub 2011 Mar 11. PMID 21397413
- [Result] Heinonen K, Raikkonen K, Pesonen AK, Andersson S, Kajantie E, Eriksson JG, Wolke D, Lano A. Behavioural symptoms of attention deficit/hyperactivity disorder in preterm and term children born small and appropriate for gestational age: a longitudinal study. BMC Pediatr. 2010 Dec 15;10:91. doi: 10.1186/1471-2431-10-91. PMID 21159164
- [Result] Schmid G, Wolke D. Preschool regulatory problems and attention-deficit/hyperactivity and cognitive deficits at school age in children born at risk: different phenotypes of dysregulation? Early Hum Dev. 2014 Aug;90(8):399-405. doi: 10.1016/j.earlhumdev.2014.05.001. Epub 2014 Jun 2. PMID 24951075
- [Result] Bauml JG, Daamen M, Meng C, Neitzel J, Scheef L, Jaekel J, Busch B, Baumann N, Bartmann P, Wolke D, Boecker H, Wohlschlager AM, Sorg C. Correspondence Between Aberrant Intrinsic Network Connectivity and Gray-Matter Volume in the Ventral Brain of Preterm Born Adults. Cereb Cortex. 2015 Nov;25(11):4135-45. doi: 10.1093/cercor/bhu133. Epub 2014 Jun 16. PMID 24935776
- [Result] Jaekel J, Wolke D. Preterm birth and dyscalculia. J Pediatr. 2014 Jun;164(6):1327-32. doi: 10.1016/j.jpeds.2014.01.069. Epub 2014 Mar 12. PMID 24630355
- [Result] Wolke D, Jaekel J, Hall J, Baumann N. Effects of sensitive parenting on the academic resilience of very preterm and very low birth weight adolescents. J Adolesc Health. 2013 Nov;53(5):642-7. doi: 10.1016/j.jadohealth.2013.06.014. Epub 2013 Jul 30. PMID 23910570
- See also: homepage — http://www.bayerische-entwicklungsstudie.de